CLINICAL TRIAL: NCT03310502
Title: Variation of Genes Controlling Carbohydrate and Lipid Metabolism
Acronym: CMgene
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Eastern Finland (Other); Kuopio University Hospital (Other); University of Turku (Other)
Responsible Party: Principal Investigator, Pirjo Nuutila, Professor, chief physician, Turku University Hospital
Other Study IDs: CMgene
Record Dates: First submitted 2017-09-21; First posted 2017-10-16 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Diabetes Mellitus, Type 2; Cardiovascular Diseases; Obesity; Insulin Resistance; Lipid Metabolism Disorders; PreDiabetes
Keywords: positron emission tomography; skeletal muscle; liver; adipose tissue; brain; genetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Obesity; Insulin Resistance; Lipid Metabolism Disorders; Prediabetic State

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of the study is to investigate genes regulating glucose and lipid metabolism in subjects whose glucose metabolism, lipid metabolism, blood flow, or body fat distribution has been measured using positron emission tomography (PET), magnetic resonance imaging (MRI), magnetic resonance spectroscopy (MRS) or computed tomography (CT) as part of their previous participation in clinical trials conducted at Turku PET Centre.

By combining information from PET, MRI, CT, proteomics, metabolomics and genetics analyses we aim to find connection between genetic variation and metabolic and cardiovascular disease.

DETAILED DESCRIPTION:
The data is collected as a separate part of the clinical imaging study protocols using a separate inform consent approved by the local ethics committee. The participation for this study consists of drawing whole blood, serum and plasma samples for genetics, proteomics and metabolomics analyses. The results from these studies are combined with baseline data from the original clinical imaging studies to find connections between genetic variation, metabolism, blood flow and body fat distribution in a cross-sectional setting.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation of studies measuring glucose metabolism, lipid metabolism, bloow flow and adiposity at Turku PET Centre

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population consists of participants of previous studies measuring glucose metabolism, lipid metabolism, bloow flow and adiposity at Turku PET Centre. Important subgroups in this study population are healthy volunteers, participants with obesity, prediabetes, type 2 diabetes or cardiovascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 2050 (Estimated)
Dates: Start 2002-04-17 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Skeletal muscle insulin sensitivity | Baseline
  Skeletal muscle glucose uptake during euglycemic-hyperinsulinemic clamp (µmol/kg tissue/min)

SECONDARY OUTCOMES:
Whole body insulin sensitivity | Baseline
  Whole body glucose uptake during euglycemic-hyperinsulinemic clamp (µmol/kg body weight/min)
Visceral adipose tissue insulin sensitivity to glucose uptake | Baseline
  Visceral adipose tissue glucose uptake during euglycemic-hyperinsulinemic clamp (µmol/kg tissue/min)
Abdominal subcutaneous adipose tissue insulin sensitivity to glucose uptake | Baseline
  Abdominal subcutaneous adipose tissue glucose uptake during euglycemic-hyperinsulinemic clamp (µmol/kg tissue/min)
Brown adipose tissue insulin sensitivity | Baseline
  Brown adipose tissue glucose uptake during euglycemic-hyperinsulinemic clamp (µmol/kg tissue/min)
Brown adipose tissue glucose uptake during cold exposure | Baseline
  Brown adipose tissue glucose uptake during cold exposure (µmol/kg tissue/min)
Insulin sensitivity of adipose tissue lipolysis | Baseline
  Plasma free fatty acid concentration during euglycemic-hyperinsulinemic clamp (mmol/l)
Myocardial insulin sensitivity | Baseline
  Myocardial glucose uptake during euglycemic-hyperinsulinemic clamp (µmol/kg tissue/min)
Liver insulin sensitivity to glucose uptake | Baseline
  Liver glucose uptake during euglycemic-hyperinsulinemic clamp (µmol/kg tissue/min)
Endogenous glucose production | Baseline
  Endogenous glucose production during euglycemic-hyperinsulinemic clamp (µmol/kg body weight/min)
Brain insulin sensitivity to glucose uptake | Baseline
  Brain glucose uptake during euglycemic-hyperinsulinemic clamp (µmol/kg tissue/min)
Abdominal subcutaneous adipose tissue mass | Baseline
  Abdominal subcutaneous adipose tissue mass (kg)
Visceral adipose tissue mass | Baseline
  Visceral adipose tissue mass (kg)
Liver fat content | Baseline
  Liver fat percentage (%)
Myocardial fatty acid uptake | Baseline
  Myocardial fatty acid uptake at fasting state (µmol/kg tissue/min)
Liver fatty acid uptake | Baseline
  Liver fatty acid uptake at fasting state (µmol/kg tissue/min)
Abdominal subcutaneous adipose tissue fatty acid uptake | Baseline
  Abdominal subcutaneous adipose tissue fatty acid uptake at fasting state (µmol/kg tissue/min)
Visceral adipose tissue fatty acid uptake | Baseline
  Visceral adipose tissue fatty acid uptake at fasting state (µmol/kg tissue/min)
Brown adipose tissue fatty acid uptake at fasting state | Baseline
  Brown adipose tissue fatty acid uptake at fasting state (µmol/kg tissue/min)
Brown adipose tissue fatty acid uptake during cold exposure | Baseline
  Brown adipose tissue fatty acid uptake at cold exposure (µmol/kg tissue/min)
Skeletal muscle fatty acid uptake | Baseline
  Skeletal muscle fatty acid uptake at fasting state (µmol/kg tissue/min)
Coronary flow reserve | Baseline
  Ratio of myocardial blood flow maximum at stress (ml/g/min) vs. myocardial blood flow at rest (ml/g/min)

CONTACTS AND LOCATIONS:
Overall Officials: Pirjo R Nuutila, MD, PhD, Principal Investigator — Turku PET centre, TurkuUH
Locations (1):
- Turku PET Centre (Turku University Hospital), Turku, Finland

IPD SHARING:
Plan to Share IPD: No
Sharing individual participant data is currently forbidden according to Finnish law.

REFERENCES:
- [Derived] Tuomola N, Rebelos E, Latva-Rasku A, Bucci M, Immonen H, Saunavaara V, Laine S, Sjoros T, Garthwaite T, Raiko JRH, Fernandes Silva L, Virtanen KA, Hannukainen JC, Ala-Korpela M, Kalliokoski KK, Heinonen IHA, Nuutila P, Honka MJ. Mildly elevated liver lipid content is characterised by reduced insulin sensitivity. JHEP Rep. 2025 Aug 6;7(11):101535. doi: 10.1016/j.jhepr.2025.101535. eCollection 2025 Nov. PMID 41113123